CLINICAL TRIAL: NCT04377334
Title: Prospective Phase II Study: MSCs in Inflammation-Resolution Programs of SARS-CoV-2 Induced ARDS
Brief Title: Mesenchymal Stem Cells (MSCs) in Inflammation-Resolution Programs of Coronavirus Disease 2019 (COVID-19) Induced Acute Respiratory Distress Syndrome (ARDS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCOVID
Record Dates: First submitted 2020-04-16; First posted 2020-05-06 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: ARDS; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC Treatment (Experimental)
  Interventions: Biological: MSC
- control (No Intervention)

INTERVENTIONS:
Biological: MSC — infusion of allogeneic bone marrow-derived human mesenchymal stem (stromal) cells
  Arms: MSC Treatment

SUMMARY:
To evaluate the safety, toxicity and immunological effects of infusion of allogeneic bone marrow-derived human mesenchymal stem (stromal) cells (MSCs) and whether this therapy has an influence on the resolution processes in ARDS patients infected with Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

ELIGIBILITY:
Inclusion Criteria:

* COVID-19-positive subject
* Horowitz index ≤ 200
* Bilateral opacities on frontal chest radiograph, and
* requirement for positive pressure ventilation via an endotracheal tube or non-invasive ventilation
* no clinical signs of left atrial hypertension detected via echocardiography, or if measured, a Pulmonary Arterial Wedge Pressure (PAOP) less than or equal to 18 mmHg.
* Subject's Age ≥ 18 years

Exclusion Criteria:

* COVID-19-negative subject
* Subject's Age < 18 years
* More than 7 days since initiation of mechanical ventilation
* Patient, surrogate or physician not committed to full intensive care support.
* Positive Pregnancy test at the time of screening.
* Patients dependent on the sponsor, investigator and their employees, as well as persons dependent on the manufacturer of the investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
lung injury score | day 10
  improvement of lung injury score (LIS), 0-16 points, severity increasing with higher points

SECONDARY OUTCOMES:
D-dimers | day 0, 1, 2, 3, 10 and 15
  D-dimers blood levels
phenotype | day 0, 1, 2, 3, 10 and 15
  distribution of phenotypes of immune cells
pro-resolving lipid mediators | day 0, 1, 2, 3, 10 and 15
  Levels of specialized pro-resolving lipid mediators within alveolar macrophages and bronchoalveolar lavage
cytokines | day 0, 1, 2, 3, 10 and 15
  Cytokine concentration within bronchoalveolar lavage and Serum prior and after MSC infusions
chemokines | day 0, 1, 2, 3, 10 and 15
  Chemokine concentration within bronchoalveolar lavage and Serum prior and after MSC infusions
Survival | day 10 and 28
  Survival at 10 days and 28 days
extubation | day 28
  Time to removal of endotracheal tube
lymphocyte subpopulations | day 0, 3, 5 and 10
  lymphocyte subpopulations in peripheral blood by flow cytometry prior and after MSC infusion (day 0,3,5,10)
SARS-CoV-2-specific antibody titers | day 0, 5 and 10
  evaluate SARS-CoV-2-specific antibody titers in the serum of patients prior and post MSC infusion.
complement molecules (C5-C9) | day 0, 5 and 10
  evaluate levels of complement molecules (C5-C9) in the serum of patients prior and post MSC infusion

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenberger, Prof., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided